CLINICAL TRIAL: NCT05840224
Title: A Phase 1 Study to Evaluate the Safety and Tolerability of GS-4528 as Monotherapy and in Combination With an Anti-PD-1 Monoclonal Antibody in Adults With Advanced Solid Tumors
Brief Title: Study of GS-4528 in Adults With Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-616-6291; 2022-502070-16 (Other: European Medicines Agency)
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor
MeSH Terms: interventions — zimberelimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1a: GS-4528 Monotherapy Dose Escalation (Experimental): Participants will receive escalating doses of GS-4528 monotherapy to determine the maximum tolerated dose.
  Interventions: Biological: GS-4528
- Phase 1a: GS-4528 Monotherapy Dose Expansion (Experimental): Participants will receive GS-4528 monotherapy at the dose determined in the escalation phase.
  Interventions: Biological: GS-4528
- Phase 1b:Dose Escalation of GS-4528 in Combination With Anti-PD-1 Monoclonal Antibody (zimberelimab) (Experimental): Participants will receive escalating doses of GS-4528 in combination with anti-PD1 monoclonal antibody (zimberelimab) to determine the maximum tolerated dose of GS-4528 as a combination therapy.
  Interventions: Biological: GS-4528; Drug: Zimberelimab

INTERVENTIONS:
Biological: GS-4528 — Administered intravenously
Drug: Zimberelimab — Administered intravenously.
  Arms: Phase 1b:Dose Escalation of GS-4528 in Combination With Anti-PD-1 Monoclonal Antibody (zimberelimab)

SUMMARY:
The goals of this clinical study are to identify if GS-4528 alone or in combination with anti-programmed cell death protein 1 (PD-1) (Anti-PD-1) Monoclonal Antibody is safe and tolerable in people with solid tumors and to identify the recommended dose of GS-4528 for further development that is safe to give to people alone or in combination with Anti-PD-1 Monoclonal Antibody.

The primary objectives of this study are:

* To assess the safety and tolerability of GS-4528 as monotherapy and in combination with Anti-PD-1 Monoclonal Antibody in participants with advanced solid tumors.
* To identify the maximum tolerated dose (MTD)/maximum administered dose (MAD) and/or the recommended Phase 2 dose (RP2D) of GS-4528 as monotherapy and in combination with Anti-PD-1 Monoclonal Antibody in participants with advanced solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented disease:

  * Phase 1a dose escalation and backfill cohorts; Phase 1b dose escalation: Individuals with histologically or cytologically confirmed advanced solid tumors who have received, been intolerant to, or been ineligible for all treatment known to confer clinical benefit or have a contraindication to receive the therapy.
  * Phase 1a dose expansion: Individuals with histologically or cytologically confirmed select indications who have received, been intolerant to, or been ineligible for all treatment known to confer clinical benefit or have a contraindication to receive the therapy.
* Eastern Cooperative Oncology Group performance status 0 or 1.
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
* Adequate organ function.
* Individuals of childbearing potential who engage in heterosexual intercourse must agree to use method(s) of contraception.
* Tissue requirements:

  * Phase 1a dose escalation, Phase 1a dose expansion, and Phase 1b dose escalation: Must provide pre-treatment adequate tumor tissue sample prior to enrolment.
  * Phase 1a backfill cohorts: Individuals must have fresh pre-treatment and on-treatment biopsy for biomarker analysis.
* Life expectancy ≥ 3 months.

Key Exclusion Criteria:

* Positive serum pregnancy test or lactating female.
* Prohibited concurrent anticancer therapy listed in the protocol.
* Any anti-cancer therapy, whether investigational or approved, within protocol specified time prior to initiation of study including: major surgery (<28 days), immunotherapy or biologic therapy (< 28 days), chemotherapy (< 21 days), targeted small molecule therapy (< 14 days or < 5 half-lives whichever is shorter), hormonal therapy or other adjunctive therapy (< 14 days) or radiotherapy (< 21 days).
* Any prior allogeneic tissue/solid organ transplantation, including allogeneic stem cell transplantation.
* Diagnosis of immunodeficiency, either primary or acquired, or systemic steroid requirement of > 10 mg of prednisone or equivalent.
* History of intolerance, hypersensitivity, or treatment discontinuation due to severe immune-related adverse events (irAEs) on prior immunotherapy.
* History of autoimmune disease or active autoimmune disease that has required systemic treatment within 2 years prior to the start of study treatment.
* Concurrent active second malignancy. Note: Individuals with a history of malignancy that have been completely treated, with no evidence of active cancer for 2 years prior to enrollment, or participants with surgically cured tumors with low risk of recurrence are allowed to enroll.
* Have known active central nervous system (CNS) metastases and/ or carcinomatous meningitis.
* Significant cardiovascular disease.
* Have active serious infection requiring antibiotics.
* Have active hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
* History of pneumonitis, interstitial lung disease, or severe radiation pneumonitis (excluding localized radiation pneumonitis).
* Symptomatic ascites or pleural effusion.
* Live vaccines within 28 days of initiation of investigational product(s).

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | First dose date up to 90 days post last dose (Up to 24 months)
Percentage of Participants Experiencing Dose Limiting Toxicities (DLTs) | Day 1 up to 4 weeks
Maximum Tolerable Dose (MTD) of GS-4528 | Day 1 up to 4 weeks

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameter: Cmax of GS-4528 as Monotherapy and in Combination With Anti-PD-1 Monoclonal Antibody | Predose on Day 1 and post dose up to end of treatment (EOT, Up to 24 months)
  Cmax is defined as the maximum observed concentration of drug.
PK parameter: Cmin of GS-4528 as Monotherapy and in Combination with Anti-PD-1 Monoclonal Antibody | Predose on Day 1 and post dose up to EOT (Up to 24 months)
  Cmin is defined as the minimum observed concentration of drug.
PK parameter: AUC of GS-4528 as Monotherapy and in Combination with Anti-PD-1 Monoclonal Antibody | Predose on Day 1 and post dose up to EOT (Up to 24 months)
  AUC is defined as the area under the concentration versus time curve.
Serum Concentrations of GS-4528 as Monotherapy and in Combination with Anti-PD-1 Monoclonal Antibody | Predose on Day 1 and post dose up to EOT (Up to 24 months)
Percentage of Participants who Develop Antidrug Antibody (ADA) Against GS-4528 | Predose on Day 1 and post dose up to 60 day follow-up (Up to 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (16):
- The University of Washington/FHCC, Seattle, Washington, United States
- Canada (2):
  - The Ottawa Hospital, Ottawa
  - University Health Network, Princess Margaret Cancer Centre, Toronto
- South Korea (3):
  - Asan Medical Center, Seoul
  - Severance Hospital, Yonsei University Health Systems, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - NEXT Oncology-Hospital Quironsalud Barcelona - Unidad de Ensayos Fase 1, Barcelona
  - Hospital Universitari Vall D'Hebron- Oncology Service, Barcelona
  - START MADRID_Hospital Universitario Fundacion Jimenez Diaz - Unidad de Ensayos Fases I, Madrid
  - START MADRID_HM Sanchinarro-CIOCC-Unidad de Ensayos Fases I, Madrid
  - Clinica Universidad de Navarra- Unidad Central de Ensayos Clinicos, Pamplona
- Taiwan (3):
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital Linkuo Branch of the Chang Gung Medical Foundation, Taoyuan District
- United Kingdom (2):
  - St Bartholomew's Hospital, London
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT05840224